CLINICAL TRIAL: NCT01325688
Title: A Phase 2 Multi-centre, Parallel Group, Open Label Study to Evaluate the Safety and Efficacy of PEP005 (Ingenol Mebutate) Gel, 0.05%, When Administered for up to Three Consecutive Days to a Superficial Basal Cell Carcinoma (sBCC) on the Trunk or Extremities
Brief Title: PEP005 Gel - Evaluation of the Safety and Efficacy of Ingenol Mebutate Gel on a Superficial Basal Cell Carcinoma on the Trunk or Extremities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-037
Record Dates: First submitted 2011-03-25; First posted 2011-03-30 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Superficial Basal Cell Carcinoma
Keywords: PEP005; Peplin; sBCC
MeSH Terms: interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): PEP005 0.05% gel applied and occluded with an aluminium disk for up to three consecutive days
  Interventions: Drug: PEP005 (ingenol mebutate) Gel, 0.05%; Device: Aluminium disk
- Group 2 (Experimental): PEP005 0.05% Gel applied and occluded with an OpSite(TM) disk up to three consecutive days
  Interventions: Drug: PEP005 (ingenol mebutate) Gel, 0.05%; Device: OpSite(TM) disk
- Group 3 (Experimental): PEP005 0.05% applied with no occlusion for up to three consecutive days
  Interventions: Drug: PEP005 (ingenol mebutate) Gel, 0.05%

INTERVENTIONS:
Drug: PEP005 (ingenol mebutate) Gel, 0.05% — PEP005 (ingenol mebutate) Gel, 0.05% for up to three consecutive days
Device: Aluminium disk
  Arms: Group 1
Device: OpSite(TM) disk
  Arms: Group 2

SUMMARY:
This study is primarily designed to investigate whether treatment, once daily for up to three consecutive days, with PEP005 (ingenol mebutate) Gel, 0.05% will be safe and tolerable in patients with superficial Basal Cell Carcinoma (sBCC) lesions on the trunk and extremities.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age
* Female patients must be of: non-childbearing potential or if of childbearing potential then have a negative serum and urine pregnancy test and using effective contraception
* Ability to provide informed consent
* primary diagnosed and histologically confirmed sBCC located on the trunk or extremities which is suitable for excision

Exclusion Criteria:

* location of the sBCC lesion within 10cm of an incompletely healed wound, on the hand or foot, on the breast of women, on the anogenital area.
* Undergone cosmetic or therapeutic procedures within 2cm of the selected treatment area in the 2 weeks prior to the screening visit.
* Use of acid-containing therapeutic products within 2 cm of the selected treatment area in the 2 weeks prior to the screening visit
* Use of topical moisturisers/creams/lotions (non-medicated/non-irritant salves are acceptable), artificial tanners or topical steroids: within 2 cm of the selected treatment area.
* Have received treatment with immunomodulators, or interferon/interferon inducers, systematic medications that suppress the immune system or UVB in the last 4 weeks
* Have undergone treatment with 5-FU, imiquimod, diclofenac or photodynamic therapy within 2 cm of the selected treatment area within 8 weeks prior to any screening visit.
* Use of systemic retinoids.
* Those who are currently participating in any other clinical trial
* Those known or suspected of not being able to comply with the requirements of the protocol
* Females who are pregnant or are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Treatment related Adverse Events, Local Skin Responses; Pigmentation and scarring | 120 days
  Number of participants with treatment related Adverse Events, change from baseline in LSR and pigmentation and scarring.

SECONDARY OUTCOMES:
Histological and clinical clearance of sBCC lesions. | 120 days
  Number of participants with histological and clinical clearance of sBCC lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Morley, Study Director — Peplin Operations
Locations (7):
- Australia (7):
  - Southderm Pty Ltd, Kogarah, New South Wales
  - St George Dermatology, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Specialist Connect, Woolloongabba, Queensland
  - Dermatology Institute of Victoria, South Yarra, Victoria
  - St John of God Dermatology, Subiaco, Western Australia
  - Burswood Dermatology, Victoria Park, Western Australia

REFERENCES:
- See also: Therapeutic Goods Administration — http://www.tga.gov.au